CLINICAL TRIAL: NCT00548964
Title: Continuation Intravenous Ketamine in Major Depressive Disorder - Modification: Lithium for Relapse Prevention
Brief Title: Continuation Ketamine in Major Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Murrough (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-1225 (002)
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine; glutamate; N-methyl-D-aspartate; treatment resistant; major depressive disorder; lithium
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Lithium; Lithium Carbonate; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine + Lithium (Experimental): All participants receive the study drug, IV ketamine, open-label
  Interventions: Drug: Lithium; Drug: Ketamine
- Ketamine + Placebo (Active Comparator): All participants receive the study drug, IV ketamine, open-label
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Lithium — 600-900mg of Li carbonate
  Other Names: Lithium Carbonate
  Arms: Ketamine + Lithium
Drug: Ketamine — 0.5mg/kg of ketamine
  Other Names: Intravenous ketamine hydrochloride

SUMMARY:
As of May 21st, 2012, the purpose of this study is to test the antidepressant effect of ketamine when given repeatedly over a period of 1 week, as well as the use of Lithium as a relapse-prevention strategy for patients with treatment-resistant depression (TRD) who respond to an initial series of ketamine infusions. Ketamine is a Food and Drug Administration approved anesthetic (a drug used to produce loss of consciousness before and during surgery). Ketamine is not approved for the treatment of major depressive disorder and is considered experimental in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 21-80 years of age;
* Female individuals who are not of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year) or using a medically accepted reliable means of contraception. Women using oral contraceptive medication for birth control must also be using a barrier contraceptive. Women of childbearing potential must also have a negative serum B-HCG at screening and at pre-infusion;
* Participants must fulfill DSM-IV criteria for Major Depression without psychotic features, based on clinical assessment by a study psychiatrist and confirmed by a structured diagnostic interview, the Structured Clinical Interview for DSM-IV TR Axis I Disorders, Patient Edition (SCID-P);
* Participants must have a history of at least one previous episode of depression prior to the current episode (recurrent MDD) or have chronic MDD (of at least two years' duration);
* Participants have not responded to two or more adequate trials of an antidepressant as determined by Antidepressant Treatment History Form (ATHF) criteria (score >=3);
* Participant scores on the IDS-C30 must be greater than or equal to 32;
* Current major depressive episode is of at least 4 weeks duration;
* Each participant must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document;
* Each participant must be able to identify a family member, physician, or friend who will participate in the Treatment Contract.

Exclusion Criteria:

* Lifetime history of psychotic features, diagnosis of schizophrenia or any other psychotic disorder, or diagnosis of bipolar disorder;
* Lifetime histories of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome;
* Current diagnosis of OCD or eating disorder (bulimia nervosa or anorexia nervosa);
* Subjects with DSM-IV drug or alcohol abuse/dependence within the preceding 2 years;
* Patients with schizotypal or antisocial personality disorder, or any clinically significant axis II disorder that would, in the investigator's judgment, preclude safe study participation;
* Patients judged clinically to be at serious and imminent suicidal or homicidal risk;
* Women who are either pregnant or nursing;
* Serious, unstable medical illnesses including hepatic, renal impairment, gastroenterologic (including gastro-esophageal reflux disease), respiratory (including obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics), cardiovascular (including ischemic heart disease and uncontrolled hypertension), endocrinologic, neurologic (including history of severe head injury), immunologic, or hematologic disease;
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
* Patients who have a positive urine toxicology for illicit substances at screening and within 24 hours of the infusion;
* Patients with one or more seizures without a clear and resolved etiology;
* Treatment with an irreversible MAOI or any other psychotropic medication within 2 weeks prior to randomization (with the exception of a stable dose of non-benzodiazepines hypnotics);
* Treatment with fluoxetine within 4 weeks prior to randomization;
* Previous recreational use of PCP or ketamine;
* Hypertension (systolic BP >160 mm Hg or diastolic BP >90 mm Hg) not controlled by diuretic or beta-blocker therapy alone or in combination;
* A blood pressure reading over 160/90 or two separate readings over 140/90 at screening or baseline visits;
* Renal impairment, as reflected by a BUN > 20 mg/dL and/or creatinin clearance of >1.3 mg/dL;
* Thyroid impairment, as reflected by a TSH > 4.2 mU/L;
* Cardiac disease, as reflected by an EKG that is abnormal and of concern for cardiac disease;
* Any anticipated change in medications that could affect fluid or salt balance, including the following antihypertensive agents: ACE inhibitor, loop diuretics, calcium channel blockers, thiazide diuretics, angiotensin II receptor blockers.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | one week

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale | one week
Quick Inventory of Depressive Symptoms | one week
Systematic Assessment for Treatment Emergent Events (SAFT) | one week
Clinical Global Impression | one week

CONTACTS AND LOCATIONS:
Overall Officials: James W Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761
- [Derived] Wan LB, Levitch CF, Perez AM, Brallier JW, Iosifescu DV, Chang LC, Foulkes A, Mathew SJ, Charney DS, Murrough JW. Ketamine safety and tolerability in clinical trials for treatment-resistant depression. J Clin Psychiatry. 2015 Mar;76(3):247-52. doi: 10.4088/JCP.13m08852. PMID 25271445
- [Derived] Murrough JW, Perez AM, Mathew SJ, Charney DS. A case of sustained remission following an acute course of ketamine in treatment-resistant depression. J Clin Psychiatry. 2011 Mar;72(3):414-5. doi: 10.4088/JCP.10l06447blu. No abstract available. PMID 21450159
- [Derived] aan het Rot M, Collins KA, Murrough JW, Perez AM, Reich DL, Charney DS, Mathew SJ. Safety and efficacy of repeated-dose intravenous ketamine for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):139-45. doi: 10.1016/j.biopsych.2009.08.038. PMID 19897179
- [Derived] Price RB, Nock MK, Charney DS, Mathew SJ. Effects of intravenous ketamine on explicit and implicit measures of suicidality in treatment-resistant depression. Biol Psychiatry. 2009 Sep 1;66(5):522-6. doi: 10.1016/j.biopsych.2009.04.029. Epub 2009 Jul 9. PMID 19545857